CLINICAL TRIAL: NCT06515717
Title: Exogenous Ketones and Behavior (ExoKet)
Brief Title: Exogenous Ketones and Behavior
Acronym: ExoKet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Responsible Party: Principal Investigator, Prof. Dr. Soyoung Q Park, Prof. Dr., German Institute of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ExoKet
Record Dates: First submitted 2024-06-19; First posted 2024-07-23 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Behavior
Keywords: ketones; human cognition; metabolism; anxiety; intervention
MeSH Terms: conditions — Behavior; Ketosis; Anxiety Disorders | interventions — formic acid 4-(3-oxobutyl)phenyl ester; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketone ester (Experimental): Participants consume a ketone ester 3x per day for 8 days.
  Interventions: Dietary Supplement: ketone ester
- Placebo containing dextrose (Placebo Comparator): Participants consume a placebo 3x per day for 8 days. The placebo is matched in calories and taste to the ketone ester.
  Interventions: Dietary Supplement: dextrose (placebo)

INTERVENTIONS:
Dietary Supplement: ketone ester — oral supplement
  Arms: ketone ester
Dietary Supplement: dextrose (placebo) — oral supplement calorie and taste matched to ketone supplement
  Arms: Placebo containing dextrose

SUMMARY:
The study will examine the effect of exogenous ketone ester on behavior and metabolism using Virtual Reality and computerizes behavioral tasks.

DETAILED DESCRIPTION:
This study investigates the effects of exogenous ketone ester on behavior, cognition, and metabolism over one week of consumption. Using a within-subjects, randomized, crossover design, participants will undergo two phases: one with the ketone ester supplement and one with a calorie- and taste-matched placebo. The study includes four lab visits: visits 1 and 3 mark the first day of each intervention, while visits 2 and 4 mark the last day. During each visit, participants will complete behavioral tasks, questionnaires, and blood tests. Additionally, participants will record their food intake via an app and collect stool samples throughout the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate
* Fluent in German
* Physically healthy. No regular medication
* No drug use 1 week prior to the study
* BMI 18-31 kg/m2

Exclusion Criteria:

* Former or current illnesses of:
* Brain or mind (including eating disorders, personality disorders, alcohol, drugs or drug dependence, neurological disorders other than occasional headache; depression or anxiety disorder excluded)
* Heart or blood circulation
* Gastro-intestinal or endocrine disorders
* Liver or kidney disorders
* Electrolyte imbalance
* Other serious past or present medical conditions (for example, metabolic syndrome, diabetes, cancer)
* Pregnancy
* Extreme athletes (>2h/day intense work-out; casual cycling or walking is ok)
* Menopause (post menopause is ok)
* Ketogenic diet, ketogenic supplement intake, intermittent fasting or calorie restricted diet during preceding 4 weeks of study participation
* Fear of blood draw

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-18 (Estimated); Primary Completion 2025-06-23 (Estimated); Study Completion 2025-06-23 (Estimated)

PRIMARY OUTCOMES:
Anxiety behavior in Virtual Reality | on day 8 of each intervention arm (visit 2 and 4)
  Using different scenes in Virtual Reality, parameters of motion behavior such as speed (measured in meters per second) and distance walked (measured in meters) will be assessed using motion tracking technology. These measurements will be combined to generate a composite score of anxiety-related motion behavior.
Risk propensity on a decision-making task | on day 8 of each intervention arm (visit 2 and 4)
  The choice (accept/reject) between a risk/gamble or safe option, based on a task paradigm by Liu et al. (2021)
Competitive confidence in a competition task | on day 8 of each intervention arm (visit 2 and 4)
  based on a task paradigm by Goette et al., 2015
Delay Discounting behavior in a computerized task | on day 1 of each intervention arm (visit 1 and 3)
  based on a task paradigm by Eisenstein et al. 2015
Performance in Dual Task | on day 1 of each intervention arm (visit 1 and 3)
  based on a task paradigm by Szameitat et al., 2002
Levels of ketones (ß-Hydroxybutyrate) | baseline, 15, 30, 60, and 90 minutes post drink-consumption on each of the 4 visits
  Blood samples
Insulin | baseline, 15, 30, 60, and 90 minutes post drink-consumption on each of the 4 visits
  Blood samples
Ghrelin | baseline and + 90 minutes post drink-consumption on each of the 4 visits
  Blood samples
Glucose Values | every 15 Minutes from visit 1 to visit 2 and again from visit 3 to visit 4
  Continuous Glucose Monitoring through sensors applied to skin
Blood Glucose | baseline, 15, 30, 60, and 90 minutes post drink-consumption on each of the 4 visits
  Blood samples
Levels of cortisol | baseline, 15, 30, 60, and 90 minutes post drink-consumption on each of the 4 visits
  Blood samples
Electrocardiogram (heart rate) | between 30 and 60 minutes post drink-consumption on each of the 4 visits
  Electrophysiological recording
Electrocardiogram (heart rate variability) | between 30 and 60 minutes post drink-consumption on each of the 4 visits
  Electrophysiological recordings
Electrodermal Activity | between 30 and 60 minutes post drink-consumption on each of the 4 visits
  Electrophysiological recordings
Subjective anxiety levels | on day 8 of each intervention arm (visit 2 and 4)
  reported by participants on visual analog scale (1-7) during Virtual Reality. 1 being no anxiety to 7 being high anxiety
Subjective stress levels | on day 8 of each intervention arm (visit 2 and 4)
  reported by participants on visual analog scale (1-7) during Virtual Reality. 1 being no stress to 7 being high stress

SECONDARY OUTCOMES:
Gut microbiome | on day 8 of each intervention arm (visit 2 and 4)
  Assessed via stool samples after each intervention
Daily food intake | 5 days of each intervention arm
  Self-reported food intake recorded via FoodApp or handwritten food diary
Trait Anxiety Questionnaire | baseline before visit 1
  Trait version of State-Trait Anxiety Inventory (STAI; Grimm et al. 2009). High scores mean high trait anxiety.
State Anxiety Questionnaire | on day 1 and 8 of each intervention arm (visit 1,2,3,4)
  State version of State-Trait Anxiety Inventory (STAI; Grimm et al. 2009). High scores mean high state anxiety.
Interoception Questionnaire | on day 8 of each intervention arm (visit 2 and 4)
  Multidimensional Assessment of Interoceptive Awareness (MAIA; Bornemann et al. 2015). High scores mean high interoceptive ability.
Depression Questionnaire | baseline, and on day 8 of each intervention arm (visit 1, 2, and 4)
  Becks Depression Inventar (BDI; Kühner et al. 2007). High scores mean high depression scores
Mood Questionnaire | on day 1 and 8 of each intervention arm (visit 1,2,3,4)
  Positive and Negative Affect Schedule (PANAS; Janke et al. 2014). High score on positive scale mean high positive mood and high scores on negative scale mean high negative mood.
Inhibition Questionnaire | baseline (visit 1)
  Behavioral Inhibition and Activation (BISBAS; Strobel et al. 2001). High scores on inhibition scale mean high inhibition and high scores on activation scale mean high activation.
Impulsivity Questionnaire | baseline (visit 1)
  Barratt Impulsiveness Scale (BIS; Barratt et al. 1965). High scores mean high impulsivity.
Social Anxiety Questionnaire | baseline, and on day 8 of each intervention arm (visit 1, 2, and 4)
  Liebowitz Social Anxiety Scale (Heimberg et al. 1999). High scores mean high scoial anxiety
Flow Questionnaire | on day 1 of each intervention arm (visit 1 and 3)
  Flow state scale (FSS; Rheinberg et al. 2002) asked after Dual Task. High scores mean more flow experience during the dual task.
Emotional Eating Questionnaire | baseline (visit 1)
  Salzburg Emotional Eating Scale (SEES; Meule et al. 2018)
Stress Eating Questionnaire | baseline (visit 1)
  Salzburg Stress Eating Scale (SSES; Meule et al. 2018)
Dominance Questionnaire | baseline, and on day 8 of each intervention arm (visit 1, 2, and 4)
  Social Dominance and Aggressive Dominance Scale (Kalma et al. 1993)
Autonomy Questionnaire | on day 8 of each intervention arm (visit 2 and 4)
  Basic Psychological Need Satisfaction and Frustration Scale (BPNSNF; Heissel et al. 2019)
Personality Questionnaire | baseline (visit 1)
  Big Five Inventory (BFI; John et al. 1991)
Chronotype Questionnaire | baseline (visit 1)
  Morningness-Eveningness Questionnaire (MEQ; Horne & Östberg, 1976)
Stress Questionnaire | baseline, and on day 8 of each intervention arm (visit 1, 2, and 4)
  Perceived Stress Questionnaire (PSQ; Fliege et al. 2001)
Subjective anxiety levels | 5 days of each intervention arm
  reported via FoodApp once per day
Subjective stress levels | 5 days of each intervention arm
  reported via FoodApp once per day

CONTACTS AND LOCATIONS:
Locations (1):
- German Institute of Human Nutrition, Potsdam, Brandenburg, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Eisenstein SA, Gredysa DM, Antenor-Dorsey JA, Green L, Arbelaez AM, Koller JM, Black KJ, Perlmutter JS, Moerlein SM, Hershey T. Correction: Insulin, Central Dopamine D2 Receptors, and Monetary Reward Discounting in Obesity. PLoS One. 2016 Jan 8;11(1):e0147063. doi: 10.1371/journal.pone.0147063. eCollection 2016. No abstract available. PMID 26744894
- [Background] Goette L, Bendahan S, Thoresen J, Hollis F, Sandi C. Stress pulls us apart: anxiety leads to differences in competitive confidence under stress. Psychoneuroendocrinology. 2015 Apr;54:115-23. doi: 10.1016/j.psyneuen.2015.01.019. Epub 2015 Feb 19. PMID 25705012
- [Background] Liu L, Artigas SO, Ulrich A, Tardu J, Mohr PNC, Wilms B, Koletzko B, Schmid SM, Park SQ. Eating to dare - Nutrition impacts human risky decision and related brain function. Neuroimage. 2021 Jun;233:117951. doi: 10.1016/j.neuroimage.2021.117951. Epub 2021 Mar 12. PMID 33722669